CLINICAL TRIAL: NCT02003001
Title: Endomyocardial Botulinum Toxin Injection Can Prevent Ventricular Arrhythmias: Pilot Study
Brief Title: Botulinum Toxin Injection to Prevent Ventricular Arrhythmias
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT_VA
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Symptomatic Ventricular Asystolia; Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Botulinum Toxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BT injection (Experimental)
  Interventions: Drug: Botulinum Toxin

INTERVENTIONS:
Drug: Botulinum Toxin

SUMMARY:
The aim of this prospective non-randomized study was to assess the efficacy and safety of endomyocardial botulinum toxin injection in left ventricle for preventing ventricular arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic ventricular arrhythmias
* drug-resistance
* unsuccessful one or more ablation procedure with future unreasonable tries

Exclusion Criteria:

* Previous heart surgery and AF ablation procedure
* Emergency CABG
* Unstable angina or heart failure
* Use antiarrhythmic drugs within 5 elimination half-lives of the drug (or within 2 months for amiodarone)
* Requiring concomitant valve surgery
* Left ventricle ejection fraction <35%
* Unwillingness to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-03 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
freedom of ventricular arrhythmias | 1 year

SECONDARY OUTCOMES:
serious adverse events | 1 year
time to recurrence of ventricular arrhythmias | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- State Research Institute of Circulation Pathology, Novosibirsk, Russia

REFERENCES:
- See also: State Research Institute of Circulation Pathology Official Site — http://meshalkin.ru